CLINICAL TRIAL: NCT01054859
Title: A PHASE I, A SINGLE-CENTRE, DOUBLE-BLIND, RANDOMIZED, PLACEBO-CONTROLLED, THREE-PERIOD, THREE-WAY CROSSOVER STUDY OF THE HEMODYNAMIC INTERACTIONS OF AVANAFIL AND ALCOHOL IN HEALTHY MALE SUBJECTS
Brief Title: A Phase I Crossover Study of the Hemodynamic Interactions of Avanafil & Alcohol in Healthy Male Subjects.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: VIVUS LLC (Industry)
Responsible Party: Wesley Day, VP Clinical Development, Vivus, Inc.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: TA-015
Record Dates: First submitted 2010-01-20; First posted 2010-01-22 (Estimated); Last update posted 2011-01-07 (Estimated); Status verified 2011-01

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — avanafil; Ethanol

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Treatment A (Experimental): 0.5 g/Kg alcohol plus 200 mg avanafil tablet
  Interventions: Drug: avanafil
- Treatment B (Active Comparator): 0.5 g/kg alcohol
  Interventions: Other: alcohol
- Treatment C (Active Comparator): 200 mg avanafil tablet
  Interventions: Drug: avanafil

INTERVENTIONS:
Drug: avanafil — 200 mg avanafil tablet QD plus 0.5 g/kg alcohol
  Arms: Treatment A
Other: alcohol — 0.5 g/kg alcohol
  Arms: Treatment B
Drug: avanafil — 200 mg avanafil tablet QD
  Arms: Treatment C

SUMMARY:
The purpose of this study is primarily to evaluate whether taking avanafil with alcohol causes the blood pressure to fall.

DETAILED DESCRIPTION:
The trial is a single-centre double-blind, randomized, placebo-controlled, three-period, three-way crossover study, in which each subject will be randomized to receive each of the following three treatments with a washout period of at least 5 days between treatments:

* Treatment A: a single oral dose of one 200 mg avanafil tablet plus an oral dose of alcohol drink mixed with fruit juice (0.5 g of absolute ethanol per kilogram of body weight).
* Treatment B: a single oral dose of one placebo tablet plus an oral dose of alcohol drink mixed with fruit juice (0.5 g of absolute ethanol per kilogram of body weight).
* Treatment C: a single oral dose of one 200 mg avanafil tablet plus an oral dose of placebo drink mixed with fruit juice.

For each treatment period, Dinamap (or DataScope) automatic measurements of supine blood pressure and pulse rate will be taken pre-dose and every 15 minutes for 4 hours post-dose. Alcohol levels using a breathalyzer will be measured at pre-dose and up to 8 hours post dose during all 3 treatments by designated unblinded personnel. Subjects should be supine for at least 5-10 minutes before the blood pressure and heart rate measurement.

ELIGIBILITY:
Inclusion Criteria:

* Adult male subjects,
* either 21 to 45 years of age,
* must be medically healthy with no clinically significant screening results.

Exclusion Criteria:

* Major exclusion criteria include: history or clinical evidence of clinically relevant cardiovascular (including thromboembolic disorders), hepatic, renal, hematological, endocrine, pulmonary, gastrointestinal, psychiatric or neurological impairment; any clinically significant laboratory abnormalities as judged by the investigator; systolic blood pressure < 90 or >150 mmHg; diastolic blood pressure < 50 or > 95 mmHg;
* allergy to or previous adverse events with PDE5 inhibitors, alcohol or their constituents; use of prescription or over-the-counter drugs that are known to interfere with metabolism by the cytochrome P450 3A4 enzyme within 30 days of Day 1 dosing (Period 1);
* use of any investigational drug within 30 days of Day 1 dosing (Period 1);
* use of any prescription or over-the-counter drugs or herbal remedies within 14 days of Day 1 dosing (Period 1);
* history of alcohol or drug abuse within 18 months, history of smoking within 6 months; positive breath alcohol, positive cotinine test or positive urine drug screen at screening or on Day -1;
* positive serology for HIV, HCV, HBsAg. Additional exclusion criteria are listed in Section 4.2.

Ages: 21 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2010-01; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
For supine systolic (SBP) and diastolic (DBP) blood pressure, the area under effect-time curve (AUEC0- t), expressed as change from baseline and the maximum decrease in blood pressure. For supine pulse rate, maximum increase in pulse rate. | 1 day

CONTACTS AND LOCATIONS:
Overall Officials: Shiyin Yee, PhD, Study Director — VIVUS LLC